CLINICAL TRIAL: NCT02773134
Title: The Early Impact of Postoperative Bracing on Pain and Quality of Life Following Posterior Instrumented Fusion for Lumbar Degenerative Conditions: A Randomized Trial
Brief Title: The Early Impact of Postoperative Bracing on Pain and Quality of Life Following Posterior Instrumented Fusion for Lumbar Degenerative Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Jean-Marc Mac-Thiong, MD, PhD, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-03-22
Record Dates: First submitted 2016-05-06; First posted 2016-05-16 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2016-05

CONDITIONS: Lumbar Degenerative Conditions
Keywords: Post-operative Bracing; Rigid Lumbosacral Orthosis; Posterior Spine Fusion; Quality of Life; Lumbar Degenerative Conditions
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brace Group (Active Comparator): Patients in the brace group will be fitted by an orthotist postoperatively and will be instructed to wear a rigid molded Lumbosacral Orthosis (LSO) full time for 8 weeks except during hygiene and wound care followed by daytime wear for another 4 weeks. All patients will start wearing the brace 48 hours after the surgery following removal of the wound drain. All braces will be molded and fitted by the same experienced orthotist affiliated with the hospital. Self-compliance to brace wear will be noted every day for 3 months by each patient on a specific form.
  Interventions: Other: Brace Group
- Control Group (Experimental): No brace prescription postoperatively. Patients in this group will be observed and results will be compared to the brace group.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Brace Group — All eligible patients will undergo a Posterior Spine Instrumented Fusion (PSIF) with the use of autologous local and iliac crest bone graft, and all pedicle screw instrumentation. A deep wound drain will be placed in all patients for 48 hours.
  All patients will complete the Oswestry Disability Index (ODI) questionnaire, the SF-12v2 General Health Survey and the Visual Analogue Scale (VAS) for back pain at baseline visit (preoperatively) and post-operatively at 6 weeks and 3 months follow up. Clinical and radiographic assessments will be performed by independent blinded observers not involved in patient care.
  Arms: Brace Group
Other: Control Group — All eligible patients will undergo a Posterior Spine Instrumented Fusion (PSIF) with the use of autologous local and iliac crest bone graft, and all pedicle screw instrumentation. A deep wound drain will be placed in all patients for 48 hours.
  Bracing will not be prescribed postoperatively for this group. All patients will the Oswestry Disability Index (ODI) questionnaire, the SF-12v2 General Health Survey and the Visual Analogue Scale (VAS) for back pain at baseline visit (pre-operatively) and post-operatively at 6 weeks and 3 months follow up. Clinical and radiographic assessments will be performed by independent blinded observers not involved in patient care.
  Arms: Control Group

SUMMARY:
Braces are commonly prescribed after posterior spinal instrumented fusion (PSIF) in patients with lumbar degenerative conditions with the aim of improving pain relief and quality of life. However, there is a lack of evidence on the indication for postoperative bracing, as surgeons choose to use braces mainly based on their experience and training.

The aim of this study is to investigate whether wearing a brace after PSIF can improve pain relief and quality of life (QOL) 6 weeks and 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with degenerative lumbar spine disease (degenerative spondylolisthesis, spinal stenosis, or degenerative disc disease);
* Patients scheduled for an elective posterior spinal fusion.

Exclusion Criteria:

* Patients with obesity (BMI > 35kg/m2).

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) score following the surgery. | Baseline, 6 weeks postoperatively, 3 months postoperatively
  The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain.

SECONDARY OUTCOMES:
Change in SF-12v2 Physical Component Score (PCS) | Baseline, 6 weeks postoperatively, 3 months postoperatively.
  SF-12v2® and SF-8™ Health Surveys measure the same eight health domains, and each survey provides psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores.
Change in SF-12v2 Mental Component Score (MCS) | Baseline, 6 weeks postoperatively, 3 months postoperatively.
  SF-12v2® Health Survey measures eight health domains and provides psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores.
Change in Visual Analog Scale (VAS) for back pain | Baseline, 6 weeks postoperatively, 3 months postoperatively.
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations.

IPD SHARING:
Plan to Share IPD: Undecided